CLINICAL TRIAL: NCT06952322
Title: Kinesiophobia in the Parents of Hemophilia Patients
Status: Completed | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Erkan KAYA, Director of Physical Medicine and Rehabilitation Clinic, Bursa City Hospital
Other Study IDs: 2025-PMR-2
Record Dates: First submitted 2025-04-18; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hemophilic Arthropathy
Keywords: Kinesiophobia; hemophilic arthropathy
MeSH Terms: conditions — Kinesiophobia | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents of Children with Hemophilia
  Interventions: Other: Questionnaire and Physical Exam
- Parents of Healthy Children
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Questionnaire results of groups will be compared.

SUMMARY:
Recurrent joint bleedings lead to the development of a debilitating arthropathy in the patients with hemophilia (PwH). This hemophilic arthropathy (HA) is characterized by chronic pain, periarticular atrophy and a limited range of motion. HA affects the perceived quality of life in the PwH. This painful situation can lead to catastrophizing thoughts that movement and physical activity will result in further pain and injury, when that painful situation is perceived as threatening. One component of this fear-model includes fear of movement, or kinesiophobia (KP). KP is defined as an irrational and disadvantaging fear of physical movement and activity resulting from feeling vulnerable to painful injury or reinjury. Patients with KP develop the belief that movements will lead to re-injury and pain. Over time, this leads to decreased physical activity, avoidance of daily tasks, functional decline, reluctance to use extremities, and in advanced stages, may result in depression and reduced quality of life. Although factors associated with KP have been examined in various diseases groups such as chronic low back pain, fibromyalgia, osteoarthritis, migraine, coronary artery disease and rheumatoid arthritis, there is limited research on KP and its predictors in PwH. To the best of our knowledge there is still no any research about effects of HA to the PwH parents' behavior differences especially regarding to KP. This study aimed to find out whether there is KP or not in the parents of patients with HA.

ELIGIBILITY:
Inclusion Criteria:

Parents of PwH and parents of healthy children were included.

Exclusion Criterias:

* Parents who failed to complete evaluation instruments
* Difficulty in understanding and writing the psychosocial evaluation questionnaires themselves
* Parents whose child has another health problem
* Parents who failed to sign the Informed Consent Document

exluded from the study.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study conducted in parents of PwH from South Marmara region and parents of healthy child from Bursa City Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Turkish version of the Tampa Scale of Kinesiophobia (TSK-19) | Day 1
  This self-administered measuring instrument consists of 19 items with a 4-point Likert scale. The score range is 11-44(a higher score indicates a greater fear of re-injury from movement).

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request data will be provided by the authors